CLINICAL TRIAL: NCT04505436
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate Efficacy, Safety and Tolerability of HM15211(Efocipegtrutide) Treatment for 12 Months in Subjects With Biopsy Confirmed NASH
Brief Title: Study to Evaluate Efficacy, Safety and Tolerability of HM15211(Efocipegtrutide) in Subjects
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM-TRIA-201
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HM15211 (Experimental)
  Interventions: Drug: HM15211
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo of HM15211

INTERVENTIONS:
Drug: HM15211 — A sterile solution of HM15211 (efocipegtrutide) contained in pre-filled syringes
  Other Names: efocipegtrutide
  Arms: HM15211
Drug: Placebo of HM15211 — A sterile, matching solution in pre-filled syringes
  Arms: Placebo

SUMMARY:
This study is a phase 2 study to Evaluate Efficacy, Safety and Tolerability of HM15211 Treatment for 12 Months in Subjects with Biopsy Confirmed NASH

ELIGIBILITY:
Inclusion Criteria:

* United States Sites: Adults ≥ 18 to ≤ 70 years.
* Korean Sites: Adults ≥ 19 to ≤ 70 years.
* BMI ≥ 18 kg/m2, with stable body weight (defined as change < 5%) by history for 3 months prior to screening or since baseline liver biopsy, whichever is earlier.
* Subjects have a diagnosis of non-cirrhotic NASH with liver fibrosis (Fibrosis stage F1-F3) confirmed by liver biopsy within 6 months of Day -7.
* MRI-PDFF performed at screening with ≥ 8% steatosis.

Exclusion Criteria:

* Subjects with a history of active or chronic liver disease, including alcoholic liver disease, viral hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, autoimmune hepatitis, Wilson's disease, hemochromatosis, alpha-1 antitrypsin deficiency, human immunodeficiency virus (HIV).
* Any history of clinically significant chronic liver disease including esophageal varices, ascites, hepatic encephalopathy, splenomegaly, or any hospitalization for treatment of chronic liver disease; or Model for End Stage Liver Disease >12.
* Recent (within 3 months of baseline biopsy) use of therapies associated with development of NAFLD (e.g., systemic corticosteroids, methotrexate, tamoxifen, aromatase inhibitors, amiodarone, or long-term use of tetracyclines).
* Type 1 diabetes subjects, or T2DM subjects on GLP-1 receptor agonist therapy, or other therapies not allowed for this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-07-27 (Estimated)

PRIMARY OUTCOMES:
pharmacodynamic (PD) effect of HM15211 | 12 months
  Proportion of subjects who achieve resolution of steatohepatitis on overall histopathological reading and no worsening of liver fibrosis

CONTACTS AND LOCATIONS:
Locations (60):
- United States (48):
  - North Alabama GI Research Center, Huntsville, Alabama
  - Synexus US - Chandler, Chandler, Arizona
  - Precision Research Institute, LLC. (PRI), Chula Vista, California
  - Fresno Clinical Research Center, Fresno, California
  - NAFLD Research Center - Altman Clinical and Translational Research Institute, La Jolla, California
  - UC Davis Health System - Midtown Ambulatory Care Center, Sacramento, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Schiff Center for Liver Diseases - University of Miami Leonard M. Miller School of Medicine(UMMSM), Miami, Florida
  - San Marcus Research Clinic, Miami Lakes, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - Ocala GI Research, Ocala, Florida
  - Synexus Clinical Research US, Inc. - Orlando, Orlando, Florida
  - Synexus Clinical Research US, Inc. - The Villages, The Villages, Florida
  - Synexus Clinical Research US, Inc, Chicago, Illinois
  - Gastroenterology Health Partners, PLLC - Southern Indiana, New Albany, Indiana
  - Kansas Medical Clinic PA (KMC) - Gastrointestinal Medical Plaza, Topeka, Kansas
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mercy Medical Center - The Institute for Digestive Health and Liver Disease, Baltimore, Maryland
  - Brigham and Women's hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Nevada Family Care & Wellness Center, Henderson, Nevada
  - Tandem Clinical Research, LLC, New York, New York
  - UNC Health Care System, Chapel Hill, North Carolina
  - Carolinas Center for Liver Disease, Carolinas HealthCare System/Atrium Health, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Lucas Research, Morehead City, North Carolina
  - Consultants for Clinical Research, Liberty Township, Ohio
  - University of Pittsburgh Medical Center (UPMC) - The Center for Liver Diseases, Pittsburgh, Pennsylvania
  - ClinSearch, Chattanooga, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Texas Liver Institute (TLI) - Texas Metabolic Center, Austin, Texas
  - The Liver Institute at Methodist Dallas, Dallas, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Liver Center of Texas, PLLC, Dallas, Texas
  - Synexus Clinical Research US, Inc, Dallas, Texas
  - Digestive Health Associates of Texas, P.A. (DHAT), Garland, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Pioneer Research Solutions Inc, Houston, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - University of Utah Health Care - UUHC - Kidney & Liver Clinic, Salt Lake City, Utah
  - Bon Secours Liver Institute of Virginia - Newport News, Newport News, Virginia
  - Virginia Commonwealth University (VCU) Medical Center, Richmond, Virginia
  - University of Washington (UW) - Harborview Medical Center (HMC) - Hepatitis and Liver Clinic, Seattle, Washington
  - Liver Institute Northwest, Seattle, Washington
- South Korea (12):
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Soonchunhyang university bucheon hospital, Bucheon-si, Gyeonggi-do
  - Natinal health insurance service Ilsan hospital, Goyang-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Seoul National University College of Medicine - Liver Research Institute, Seoul, Seoul
  - Severance Hospital, Seoul, Seoul
  - SMG-SNU Boramae Medical Center, Seoul, Seoul
  - EWHA Womans University Mokdong Hospital, Seoul, Seoul
  - Korea University Guro Hospital, Seoul, Seoul
  - Eunpyeong St. Mary Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No